CLINICAL TRIAL: NCT02354469
Title: The Effects of Head Trauma on Biological Markers and Neurologic Function in Collegiate Athletes: a Prospective Investigation
Brief Title: The Effects of Head Trauma on Collegiate Athletes
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Harvard University (Other); Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other); Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, David R Howell, Assistant Professor, University of Colorado, Denver
Other Study IDs: IRB-P00016469
Record Dates: First submitted 2015-01-29; First posted 2015-02-03 (Estimated); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Cerebral Concussion; Brain Injuries
Keywords: TBI; Mild Traumatic Brain Injury; Post-Concussion Syndrome; Recovery of Function; Motor Activity; Diffusion Tensor Imaging; Neural Injury; Biomarkers
MeSH Terms: conditions — Brain Concussion; Brain Injuries; Post-Concussion Syndrome; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine and blood samples will be acquired and stored in a biorepository.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Contact/Collision Sport Athletes: Collegiate athletes who participate in contact or collision sports will be assessed on a comprehensive battery of tests during pre-season and post-season assessments.
- Non-contact Sport Athletes: Collegiate athletes who participate in non-contact sports will be assessed on a comprehensive battery of tests during pre-season and post-season assessments.
- Post-Concussion: Collegiate athletes who sustain a concussion will be assessed on a comprehensive battery of tests from the time of injury and incrementally throughout the following year post-injury.
- Healthy Control: Collegiate athletes who do not sustain a concussion but match the demographic profile of an individual enrolled as a post-concussion subject, will be assessed on the same tests and in a similar timeline as post-concussion subjects.

SUMMARY:
Recently, researchers and clinicians have examined many different forms of concussion testing aimed to assess if a brain injury has occurred and to what degree it affects the individual being tested. Due to the multifaceted and complex presentation of concussive injuries and the unknown effects of repeated head trauma, it is unlikely that a single test of physiological or behavioral function will reflect the full range of injury-related damages from a concussive event or from a series of cumulative head traumas, as well as the injury response within brain tissue. However, by combining a variety of objective assessments which may detect structural and functional alterations following head trauma into a single study, a clearer understanding of the multi-faceted presentation resulting from head trauma may be identified. The identification of biomarkers and the utilization of objective and clinically feasible tools will provide a method to assess three domains across multiple systems affected by head trauma: 1) the prognostic value of initial concussion assessments to identify injury severity and factors responsible for prolonged recovery, 2) the temporal window of recovery and potential vulnerability of brain tissue post-injury, and 3) the long-term alterations associated with repeated head trauma exposure.

DETAILED DESCRIPTION:
Student athletes from contact and collision sports, as well as non-contact sports, will complete a comprehensive assessment of neurological and behavioral function before and after a season of participation. Additionally, those who sustain a concussion will undergo a post-injury testing timeline where they are assessed within 5 days of injury and again at the following time points: 3-4 weeks, 3 months, 6 months, and 1 year post-injury. Each individual who completes testing as a concussion subject will be matched with a healthy control subject by height, weight, age, sport, and position, and each control subject will complete the same protocol in similar time increments as subjects with concussion.

Through this study design, we hypothesize that we will be able to detect objective deficits resulting from concussion within one week of injury and determine the feasibility and added value of a comprehensive neurological and behavioral testing battery through a comparison of metrics between injured and healthy collegiate student athletes. Additionally, we hypothesize that for athletes who do not sustain a concussion, decrements between the pre-season and post-season time points will be greater in those who participate in collision/contact sports in comparison to those who participate in non-contact sports. Thus, outcomes from this study will enhance the understanding of the pathophysiology of concussion through a rigorous laboratory testing component, but with simultaneous direct translation to clinical implementation through the use of a highly-feasible clinical testing paradigm that possesses potential for ubiquitous and widespread use throughout sports medicine practices.

ELIGIBILITY:
Inclusion Criteria:

1. Participation on a Harvard University varsity athletic team
2. Medically cleared to participate in sport, as determined by Harvard medical staff
3. Diagnosed with concussion by Harvard medical staff, and agreement to participate in the post-injury component of the study within five days of injury (post-concussion group)
4. No diagnosed concussion within the previous year of evaluation (control group)

Exclusion Criteria:

1. A history of epilepsy, prior seizure, or any previous abnormal EEG finding or abnormal brain imaging (CT or MRI) finding, as reported by the patient.
2. Any pre-existing neurological disorder, including but not limited to stroke, intracranial hemorrhage, any movement disorder, and cerebral palsy.
3. Any currently active psychiatric condition, including specifically major depression, bipolar disorder or schizophrenia. A history of a psychiatric condition but no ongoing psychiatric episode (e.g. not currently undergoing treatment for a major depressive episode) would not be an exclusion.
4. Any unstable medical condition
5. For the transcranial Doppler ultrasound component of the study only, subjects with infection, history of seizure, cardioactive drug participation, presence of deep vein thrombosis, cervical injury (structural or vascular), gross motor deficits, or skull fractures will be excluded.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects will be comprised of active members of various varsity teams at Harvard University.
Sampling Method: Non-Probability Sample
Enrollment: 437 (Actual)
Dates: Start 2015-08; Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Dynamic Balance Control | 1 year
  For balance control measures, the primary data will come from accelerometers placed on specific anatomical landmarks to assess whole body movement. Peak accelerations and velocities of an estimated center-of-mass during gait under single-task and dual-task conditions will identify how divided attention tasks affect whole body balance control.

SECONDARY OUTCOMES:
Cognitive Function | 1 year
  Concussion-Rapid Assessment Module, simple and choice reaction times, Trail Making Tests A and B, Balance Error Scoring System, and static and dynamic visual acuity will be assessed.
EEG signals | 1 year
  We plan to examine a variety of conventional EEG measures including resting-state power and functional connectivity, as well as task-related evoked potentials, functional connectivity changes, and event-related spectral perturbation.
Blood and Urine samples | 1 year
  We will primarily investigate previously documented markers of neuronal integrity GFAP, UCH-L1, and SB100 (blood) and levels of protein concentration in urine
Neuroimaging | 1 year
  Primary measures will include: gross and regional volumes of brain structures, water molecule diffusion (axial diffusivity, fractional anisotropy, radial diffusivity, and mean diffusivity), and neurochemical imaging (levels of NAA, Cr, Cho, Glu, GSH, and MI).

CONTACTS AND LOCATIONS:
Overall Officials: William P Meehan III, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Howell DR, Brilliant A, Berkstresser B, Wang F, Fraser J, Meehan WP 3rd. The Association between Dual-Task Gait after Concussion and Prolonged Symptom Duration. J Neurotrauma. 2017 Dec 1;34(23):3288-3294. doi: 10.1089/neu.2017.5191. Epub 2017 Oct 16. PMID 28895490
- [Background] Howell DR, Stillman A, Buckley TA, Berkstresser B, Wang F, Meehan WP 3rd. The utility of instrumented dual-task gait and tablet-based neurocognitive measurements after concussion. J Sci Med Sport. 2018 Apr;21(4):358-362. doi: 10.1016/j.jsams.2017.08.004. Epub 2017 Aug 16. PMID 28919121
- [Background] Howell DR, Oldham JR, DiFabio M, Vallabhajosula S, Hall EE, Ketcham CJ, Meehan WP 3rd, Buckley TA. Single-Task and Dual-Task Gait Among Collegiate Athletes of Different Sport Classifications: Implications for Concussion Management. J Appl Biomech. 2017 Feb;33(1):24-31. doi: 10.1123/jab.2015-0323. Epub 2016 Oct 5. PMID 27705076
- [Background] Howell DR, Buckley TA, Berkstresser B, Wang F, Meehan WP 3rd. Identification of Post-Concussion Dual-Task Gait Abnormalities Using Normative Reference Values. J Appl Biomech. 2019 Aug 1;35(4):290-296. doi: 10.1123/jab.2018-0454. Epub 2019 May 29. PMID 31141425
- [Background] Howell DR, Buckley TA, Lynall RC, Meehan WP 3rd. Worsening Dual-Task Gait Costs after Concussion and their Association with Subsequent Sport-Related Injury. J Neurotrauma. 2018 Jul 15;35(14):1630-1636. doi: 10.1089/neu.2017.5570. Epub 2018 May 3. PMID 29490564
- [Derived] Daisy CC, Varinos S, Howell DR, Kaplan K, Mannix R, Meehan WP, Wang F, Berkstresser B, Lee RS, Froehlich JW, Zurakowski D, Moses MA. Proteomic Discovery of Noninvasive Biomarkers Associated With Sport-Related Concussions. Neurology. 2022 Jan 11;98(2):e186-e198. doi: 10.1212/WNL.0000000000013001. Epub 2021 Oct 21. PMID 34675105